CLINICAL TRIAL: NCT01431443
Title: Consumption of Chocolate in Pregnant Women at High Risk for Preeclampsia.
Brief Title: Consumption of Chocolate in Pregnant Women.
Acronym: CHOCENTA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IC096501
Record Dates: First submitted 2011-05-02; First posted 2011-09-09 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Preeclampsia
Keywords: Randomized double blind trial; Cocoa flavonoids; Endothelial function; Blood pressure; Pregnant women; Preeclampsia; Uterine artery flow; Pulsatility index
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dark chocolate (Experimental)
  Interventions: Other: Flavanol-rich chocolate
- Placebo chocolate (Placebo Comparator): Placebo intervention
  Interventions: Other: Placebo Chocolate

INTERVENTIONS:
Other: Flavanol-rich chocolate — The aim of this study is to evaluate the beneficial effect of dark chocolate consumption through the activity of flavanols on the endothelial function and blood pressure regulation, in acute (after 3 hours) and chronic effect (12 weeks), among pregnant women at high risk for preeclampsia.
  Arms: Dark chocolate
Other: Placebo Chocolate — Placebo intervention
  Other Names: Flavanol and theobromine-free chocolate
  Arms: Placebo chocolate

SUMMARY:
The purpose of this study is to investigate the acute and chronic effect of consumption of flavanol-rich chocolate on endothelium function in pregnant women at high risk for preeclampsia.

DETAILED DESCRIPTION:
Although numerous strategies have been studied, no effective prevention or treatment of preeclampsia is yet available for pregnant women. This is surprising considering the growing body of literature that supports the hypothesis of a beneficial effect of dark chocolate consumption through the activity of flavanols on the endothelial function and blood pressure regulation, to find any clinical data among pregnant women with preeclampsia.

The primary objective of the trial is to investigate the acute and chronic effect of consumption of flavanol-rich chocolate on endothelial function in pregnant women at high risk of preeclampsia. This 12-week efficacy study will permit us to verify the sustainability of the effect of daily intake of flavanol-rich chocolate intake.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between the ages of 18 and 40 years.
* Presence of uterine diastolic notches measured by uterine artery Doppler between 10 and 14 weeks.

Exclusion Criteria:

* Hypertension requiring medication.
* Currently or previously use of medications interfering with glucose or lipids metabolism.
* Use of supplements or natural health products that interfere with blood pressure.
* Consumption of 1 or more alcohol drink per day.
* Allergy or intolerance to nuts or chocolate.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2011-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Changes in endothelial function | within the first 12 weeks of chocolate intake

SECONDARY OUTCOMES:
Doppler of uterine arteries | within the first 12 weeks of chocolate intake
Blood pressure | within the first 12 weeks of chocolate intake
Plasma biomarker of endothelium function | within the first 12 weeks of chocolate intake
Plasma biomarker of chocolate intake | within the first 12 weeks of chocolate intake
  ng\ml plasma

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Dodin, MD, Principal Investigator — Laval University
Locations (1):
- Laval University, Department of Medicine, Institut des nutraceutiques et des aliments fonctionnels., Québec, Quebec, Canada